CLINICAL TRIAL: NCT06646653
Title: Feasibility Clinical Study of the Alma System in Treating Primary Postpartum Hemorrhage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ResQ Medical Ltd (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD-01-002-PR
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Postpartum Haemorrhage (PPH); PPH; Postpartum Hemorrhage (Primary)
Keywords: Alma System; postpartum hemorrhage; pph
MeSH Terms: conditions — Postpartum Hemorrhage; Familial Primary Pulmonary Hypertension

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized, feasibility pilot study of 10 women with vaginal or caesarean deliveries in a hospital setting who failed first-line interventions for postpartum hemorrhage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participant group (Experimental): Woman who developed PPH after vaginal or caesarean delivery and first line interventions have been attempted and failed, and to which the Alma System was applied
  Interventions: Device: Alma System

INTERVENTIONS:
Device: Alma System — Subjects diagnosed with postpartum hemorrhage will receive the Alma System. This system comprises a soft silicone cylindrical device placed within the uterus. Gentle suction is applied, prompting the uterus to contract and reduce in size. This contraction compresses the blood vessels, halting the bleeding.
  Other Names: Obstetric-gynecologic specialized manual instrument; Vacuum induced heamorrhage control

SUMMARY:
Feasibility clinical study of the Alma System in treating primary postpartum hemorrhage (PPH).

DETAILED DESCRIPTION:
10 subjects, first in woman trial with ethics committee oversight. Women who experienced postpartum hemorrhage will be treated with the Alma System, which aims to rapidly reduce or stop the bleeding by targeting the primary cause: uterine atony.

The primary objective is to verify the safety of the Alma System in humans by: 1. Ensuring the absence of serious adverse events (SAEs) related to the use of the Alma System during and after the procedure. 2. Evaluating any observable damage to the uterus, cervix, or vagina due to the use of the Alma System. 3. Evaluating the occurrence of uterine inversion or folding during the use of the Alma System.

The secondary objectives include evaluating: 1. The ability to easily place the Alma System trans-vaginally. 2. The ability to connect the Alma System to a vacuum source and maintain the desired negative pressure. 3. The ability of the Alma System to contract the uterus to a level that reduces or stops blood loss and avoids further non-surgical and surgical intervention. 4. The time from insertion and start of negative pressure to a visible reduction in blood loss.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Female, 18 years of age or older at time of consent.
2. Subject or her legally authorized representative is able to understand and provide consent to participate in the clinical investigation.
3. Subjects who present with an atonic uterus for at least 10 minutes after expulsion of placenta with failure to obtain contraction and/or Subjects who have lost blood post-vaginal delivery > = 500 ml and lost blood post-cesarian delivery > = 1000 ml and according to the Investigator's judgment, require an intervention.
4. Failed first-line intervention of uterotonics and uterine massage/bimanual uterine massage to stop bleeding.

Exclusion Criteria:

1. Subjects who do not provide informed consent to participate in the clinical investigation.
2. Subjects who deliver at a uterus size < 34 weeks.
3. Subjects who have lost > 1000 ml of blood for vaginal birth and > 2000 ml for caesarian delivery.
4. Subjects who have abnormal PT, PTT and INR.
5. Subjects who present with retained placenta, uterine lacerations, or for any other conditions outside of atonic post-partum hemorrhage.
6. PPH that the investigator determines to require more aggressive treatment, including any of the following:

   * Hysterectomy;
   * B-lynch suture;
   * Uterine artery embolization or ligation;
   * Hypogastric ligation;
   * Known uterine anomaly;
   * Ongoing intrauterine pregnancy.
7. Placental abnormality including any of the following:

   * Known placenta accreta;
   * Retained placenta with known risk factors for placenta accreta (e.g., history of prior uterine surgery, including prior c-section and placenta previa);
   * Retained placenta without easy manual removal.
8. Known uterine rupture
9. Unresolved uterine inversion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-14 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Rate of related SAEs | 6 weeks
  Rate of device related SAEs up to six weeks following device treatment
Rate of Damage to Cervix, Uterus or Vagina | Procedure
  Rate of any observable damage to cervix, uterus or vagina during or immediately after device procedure
Rate of Occurrence of Uterine Inversion or Folding | Procedure
  Rate of occurrence of uterine inversion or folding during or immediately after device procedure

SECONDARY OUTCOMES:
User Feedback on Connection to Vacuum | Procedure
  Rate of positive user feedback on connection to vacuum and maintenance of desired negative pressure
Rate of Uterine Contraction | Procedure
  Rate of uterine contraction to a level that reduces or stops blood flow
Time to Visible Reduction in Blood Flow | Procedure
  Time from insertion and start of negative pressure to visible reduction in blood flow
User Feedback on Placement of Alma | Procedure
  Rate of positive user feedback on device placement transvaginally

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinical Hospital of Mostar, Mostar, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: Undecided